CLINICAL TRIAL: NCT01449604
Title: Randomized Comparison of Steretotactic Radiosurgery and Hypofractionated Steretotactic Radiotherapy in the Treatment of Vestibular Schwannoma
Brief Title: Stereotactic Radiation in Vestibular Schwannoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Putipun Puataweepong, Assistant professor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAMART0111
Record Dates: First submitted 2011-10-02; First posted 2011-10-10 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Vestibular Schwannoma
Keywords: Stereotactic radiotherapy; SRS; SRT; vestibular schwannoma
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- stereotactic radiosurgery (Active Comparator): Radio surgery single fraction 12 Gy
  Interventions: Radiation: stereotactic radiosurgery
- stereotactic radiotherapy (Active Comparator): Stereotactic radiotherapy hypo fraction 18 Gy in 3 fraction
  Interventions: Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: stereotactic radiotherapy — Stereotactic radiotherapy, hypofraction using 18 Gray in 3 fractions
  Arms: stereotactic radiotherapy
Radiation: stereotactic radiosurgery — Radio surgery 12 Gy
  Other Names: SRS
  Arms: stereotactic radiosurgery

SUMMARY:
The purpose of this study is to determine whether stereotactic radiosurgery (SRS)and stereotactic radiotherapy (SRT)are effective in the treatment of vestibular schwannoma (VS).

DETAILED DESCRIPTION:
Vestibular schwannomas (VSs) are slow-growing tumors of the myelin-forming cells that cover cranial nerve VIII.The treatment options for patients with VSs include active observation, surgical management, and radiotherapy. However, the optimal treatment choice remain controversial.

Over the past 10 years, there has been rapid progress in the application of stereotactic radiotherapy to the treatment of VSs. The stereotactic radiotherapy program includes single fraction radiosurgery (SRS) and hypofraction stereotactic radiotherapy (HSRT) are commonly used for VSs treatment. Since SRS and SRT techniques differ significantly enough to raise questions of therapeutic advantage and until now, there is no prospective, randomized study comparing the outcomes for patients treated using both radiotherapy techniques. We designed the first prospective randomized protocol to compare SRS and SRT for answer this question.

ELIGIBILITY:
Inclusion Criteria:

* vestibular schwannoma tumor size not more than 3 cm.

Exclusion Criteria:

* NF 2 patient
* underlying cerebrovascular disease
* tumor compress and efface brain stem ( Koos 4)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
audiogram | two year
  change from baseline audiogram at 6 months,1 year and 2 year

SECONDARY OUTCOMES:
number of participant with adverse event | 2 year
  the new number of adverse event after radiation at 6 month,1 and 2 year
tumor size | 2 year
  change in tumor size at 6 month, 1 year and 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Putipun Puataweepong, M.D., Principal Investigator — Ramathibodi Hospital